CLINICAL TRIAL: NCT01572883
Title: Effect of Concomitant Radiotherapy and Trastuzumab on Cardiotoxicity of Patients Treated for Early Breast Cancer
Status: Completed | Type: Observational
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: eHER2-TM
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Breast Cancer
Keywords: adjuvant treatment with Radiotherapy and trastuzumab
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether concomitant radiotherapy and trastuzumab (patients treated for early breast cancer) is really safe for the heart even years after treatment and if the investigators should use these two treatments concomitantly without additional harm.

DETAILED DESCRIPTION:
The investigators know from the studies, that were already published, that for HER2 positive early breast cancer patients in adjuvant treatment concomitant radiotherapy and trastuzumab is safe during the treatment. But there is no study with long term results of cardial function, especially combination of Left ventricular ejection fraction (LVEF) and NT-proBNP.

ELIGIBILITY:
Inclusion Criteria:

* Early breast cancer patients,treated adjuvantly with radiotherapy of the operated breast or thoracic wall and treated concomitantly with trastuzumab.
* Reviewed many months after treatment, without recurrence of disease.

Exclusion Criteria:

* Recurrence of disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: breast cancer patients treated in Institut of Oncology Ljubljana,slovenia since year 2005.
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2011-12; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
difference in LVEF (Left Ventricular Ejection Fraction) | from one to six years from adjuvant radiotherapy for early breast cancer
  we will compare LVEF (LVEF 1) measured before treatment with adjuvant Trastuzumab and concomitant Radiotherapy of breast/thoracic wall with LVEF (LVEF 2) measured at follow up (after adjuvant treatment) outpatient examination. We will then compare the difference in LVEF (LVEF 2-LVEF 1) measured in patients treated for left breast cancer with the difference in LVEF (LVEF 2-LVEF 1) measured in patients treated for right breast cancer

SECONDARY OUTCOMES:
occurrence of cardiovascular events over time in both groups (RT for left/right breast) | from 6 months to five years after adjuvant therapy with trastuzumab
  occurrence of cardiovascular events over time in both groups (irradiated left / right breast) will be showed by the method of Kaplan-Meier. Groups will be compared with the log rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Marinko, MD, Principal Investigator — Institute of Oncology Ljubljana
Locations (1):
- Institut of oncology Ljubljana, Ljubljana, Slovenia